



#### **PROTOCOL COVER PAGE**

**PROTOCOL NAME:** Outcome of a lecture before vs after simulation-based education on pediatric status epileptics: A randomized controlled pilot trial

#### PRINCIPAL INVESTIGATOR:

Dr. Melissa Chan BC Children's Hospital

4500 Oak St. Vancouver, BC. V6H 3N1

#### **Co-Investigators:**

Dr. John Ramsay BC Children's Hospital 4500 Oak St.

Vancouver, BC.

V6H 3N1

Phone: 613-223-4513

Email: ramsay.s.john@gmail.com

Dr. Jonathan Duff

Stollery Children's Hospital

8440 112 St. NW Edmonton, AB.

T6G 2B7

Funded By: Not applicable

**Current Protocol Version: Protocol Version #0.1, Aug 16, 2023** 

**H Number:** H22-03760





#### 1 Protocol Summary

#### 1.1 Synopsis

**Title:** Comparing teaching before vs after simulation education on pediatric status epileptics: A randomized controlled trial

**Study Description:** The study will test whether simulation preceding didactic teaching leads to improved knowledge and performance retention compared to a didactic lecture proceeding simulation. Participants will be randomized to one of two different groups: 1) didactic teaching followed by simulation or 2) simulation then didactic teaching.

#### **Primary Outcomes**:

- 1. Resuscitation performance retention score 3 months post-initial training Secondary Outcomes:
  - 2. Knowledge assessment 3 months post-initial training
  - 3. Learner satisfaction

#### **Hypothesis:**

1. Didactic teaching after simulation-based training will be more effective in maintaining retention of knowledge and skills in the management of pediatric status epilepticus compared to didactic teaching prior to simulation

**Study Population:** Second year medical students from the University of British Columbia – Vancouver Campus

**Description of Sites:** The intervention will take place at BC Children's Hospital Simulation Centre with trained facilitators and high-realism simulation equipment.

**Description of Study Intervention:** One arm of the study will receive a 60-minute lecture on pediatric status epilepticus management and then complete a simulation scenario immediately after. The second arm will complete a simulation scenario on pediatric status epilepticus without knowing the topic beforehand and will complete a 60-minute lecture immediately after the simulation session. Both groups will complete a knowledge test directly after the intervention. Both groups will be reassessed in three months with a repeat simulation scenario on pediatric status epilepticus and repeat knowledge test.

**Study Duration** The study will enroll participants for 2 months and then complete the educational intervention over 3 months.

**Participant Duration:** The participants will participate in one 60-minute lecture and two ten-minute simulation sessions and one focused 15 minute debrief over the course of four months' time.



Figure 1: Flow of participants through the research project





#### 2 Introduction

#### 2.1 Background Information & Rationale

Simulation is a revolutionary tool in medical education and specifically pediatrics with the rarity of lifethreatening situations. It provides learners with the opportunity to practice high-stress crucial medical scenarios in a safe and supportive environment where mistakes are instead valuable teaching for future experiences. Simulation has been shown to be an effective teaching method in medical education however how best to optimize retention and patient outcomes remains unclear<sup>1–3</sup>. Medical education interventions are typically evaluated at one stage of Kirkpatrick's framework for learning which include reaction (level 1), learning (level 2), behavior (level 3) and results (Level 4)<sup>4</sup>. Patient outcomes remains the strongest measure however is difficulty to effectively design projects to show this<sup>5,6</sup>. In pediatrics procedures and adult ACLS retention of knowledge and skills have been shown to decline by as early as 3-months' time in two systematic reviews<sup>7,8</sup>. In our assessment, it remains unclear what the best method of teaching associated with simulation is and when the best time to facilitate this teaching to improve retention for medical expert knowledge and resuscitation performance.

Pre-simulation assignments may be an effective way to prime participants for learning in simulation. Different methods including reading, written assignments, plan of care mapping, pre-quizzes, scenario demonstration, virtual reality, lectures and online games have been described<sup>9–16</sup>. No method has been identified as superior<sup>17,18</sup>. Pre-simulation preparation was felt to improved learning in one systematic review however the strength of the evidence was weak and primarily level 1 and 2 outcomes were assessed<sup>17,19</sup>. There remains contention in the literature with one study finding adding simulation to a flipped classroom teaching model improving 3-month retention though multiple studies examining a flipped classroom model in rapid-cycle deliberate practice models found no improvement<sup>11,20,21</sup>. New evidence suggests there may be better immediate knowledge gain from simulation preceding didactic teaching compared to didactic teaching before simulation<sup>22,23</sup>. For procedural skills it has been shown the practical sessions before theory-based lectures resulted in increased skill and knowledge retention at one month for transesophageal echocardiography<sup>24</sup>.

Pediatric seizure is a common acute care pediatric scenario with numerous published simulation scenarios<sup>25–27</sup> and evaluation rubrics available as well as multiple high-quality national pediatric status epilepticus management algorithms available<sup>28,29</sup>. The effect of pre and post simulation teaching remains debated in medical education literature as well as the ongoing concern of knowledge and performance degradation. This study aims to investigate the effect of pre and post teaching on knowledge degradation, and how to best optimize knowledge retention to improve medical education and theorized patient care. The specific objectives are to assess whether teaching before or after a simulation leads to medical students' improved knowledge and resuscitation performance retention at two to fourth months post educational intervention for managing pediatric status epilepticus.





#### 2.2 Risk/Benefit Assessment

#### 2.2.1 Known Potential Risks

As this is a medical education study there are minimal risks to the participants. The participation in simulation could cause increased stress to the learner but this will be minimized with structured pre-brief and debrief sessions.

#### 2.2.2 Known Potential Benefits

The participants will benefit from two simulation teaching sessions with a trained simulation expert and FRPC certified pediatric emergency medicine physician. They will also receive an additional lecture providing them with didactic teaching on status epilepticus.

### 3 Objectives

The primary objective is to assess the resuscitation performance retention difference between the two educational intervention arms at two to four months following teaching.

The secondary objectives are to assess the difference in knowledge between both study groups immediately after and two to four months after the educational intervention. In addition, we will measure the comfort of learners performing the initial simulation scenario.

#### 3.1 Outcome Measures

The primary outcome will be the resuscitation performance retention assessed using the post-teaching the final global rating scale score (1-7 performance score) for medical management and flow during each simulation as well as the following "time-to" metrics; glucose check, IV access, chemistry panel order, first-line anti-epileptic administration<sup>30</sup>, second line anti-epileptic administration. This will be adjusted for baseline score.

The secondary outcome measures for knowledge retention assessment will be the post-teaching knowledge test score assessed on a 15 Question MCQ test administered at the final assessment adjusted for the baseline score.

Comfort/Confidence will be assessed using the change in Likert scale item after each simulation and debrief.

## 4 Study Population

#### 4.1. Inclusion Criteria

1. Second year medical students at the University of British Columbia – Vancouver Campus

#### 4.2 Expected Duration of Subject Participation

A participant will already be expected to attend a 60 min teaching session on status epilepticus. They will also be required to participate in two 10-25 min simulation sessions which will include a 10-minute simulation and 15 debrief for the first and only a 10-minute simulation the second time.





#### 4.3 Recruitment and Retention

The study participants will be recruited from the second-year medical student cohort at the University of British Columbia Vancouver campus. A medical student assisting in the research project will be the primary point for recruiting medical students and will post regularly in medical student communication channels including but not limited to Slack, Facebook and word of mouth. The participants names and contact information will be saved at this stage to allow for scheduling of the simulation and teaching sessions.

The consent form will be emailed to participants to complete prior to participation and researchers will be available for questions.

#### 5 Study Design

#### 5.1 Overall Design

This is a parallel randomized control trial in medical education that will be conducted at the BC Children's Hospital. The participants will be masked to the other arm of the intervention and the outcome measures of the study.

#### 5.2 Data Collection

The simulation sessions will be recorded to ensure accuracy in time to intervention recordings and global rating scales. Two experienced pediatric acute care specialists with simulation experience masked from the intervention arms will review the videos and determine the global rating scale for each simulation and they will review videos for the "time to metrics". Time zero will be immediately after the scenario description is completed.

The knowledge tests and anxiety/confidence assessment will be completed using a redcap-hosted survey. Basic demographic information including age, previous experience with simulation and a background in ED nursing or EMS will also be collected using a demographic survey. The names and contact information will not linked to the demographic or simulation information. This survey can be found in appendix A.

#### 5.3 Didactic Lecture and Simulation Development:

The lecture and two simulation scenarios were developed by the primary researcher, a first-year pediatric emergency medicine fellow with guidance from the principal investigators, a pediatric intensivist and pediatric emergency medicine specialist who both have expertise in simulation and curriculum development. Both the lecture and simulations were peer-reviewed by a pediatric emergency medicine specialist with simulation expertise who was not involved with research project.

The lecture was developed using existing pediatric seizure management guidelines from Trekk and the Canadian Pediatric Society<sup>28,29</sup>. The lecture learning objectives mirrored the research outcome measures and focused on acute management of pediatric seizures with supporting discussions on possible etiologies. It did not discuss crisis-resource management skills, long-term management or prognosis of seizures or other acute pediatric scenarios. The lecture can be found in PDF form in Appendix B.





The simulation scenarios were developed using published pediatric seizure scenarios as a baseline and set at a level appropriate for trainees with limited clinical experience. The pediatric status epilepticus scenarios can be found in appendix C.

#### 5.4 Study Protocol:

The participants will be randomized into two groups: Lecture-> Simulation -> Evaluation Simulation(LS) and Simulation->Lecture -> Evaluation Simulation (SL) using blocked randomization with varied block size. The randomization allocation sequence will be completed by RedCap and the researchers will be masked to this.

The LS group will complete the 60-minute focused lecture immediately prior to their initial simulation. The SL group will complete the 60-minute focused lecture immediately after their initial simulation. The LS group will complete a pre-intervention knowledge test prior to the lecture and the SL group will complete a knowledge test prior to the initial simulation.

Both groups will complete the initial simulation in groups of 3-4 with one member acting as the leader and others acting as team members. The simulation will last for 10 minutes followed by a structure debrief using the +/delta method lasting up to 20 minutes. The debrief will be completed by a pediatric emergency medicine specialist with experience in leading simulation debrief. The leader of the group will be recorded for later subgroup analysis.

Every individual will complete a second evaluatory simulation 3 months after the initial simulation to evaluate the primary outcome of resuscitation performance retention. Each participant will act as the simulation leader with two actors who will function as a highly trained nurse and second physician but will not provide advice. The simulation will be videotaped. The participants will also complete a knowledge test prior after the second simulation.

Simulation videos will be reviewed as per the above data collection method to determine outcome measures. The simulations will be completed in the BCCH simulation center with a trained pediatric simulation expert and simulation facilitator. A high-fidelity mannequin will be used. It can seize and has appreciable chest rise and breath sounds. The participants will be instructed to assume all medications requested are drawn up in a syringe to the dose desired in the medication tray to decrease variability in time to metrics from difficulty in drawing up medications.

#### 6 Statistical Consideration

## **6.1** Sample Size Determination:

The one paper assessing knowledge and skill retention comparing SL and LS structured teaching found a 13.42% difference in skill performance on transesophageal echocardiography<sup>24</sup> with the following means and std; LS group 71.90 (18.59) and SL group 85.32(15.63). Using a sample size calculator estimates a sample size of 60 with an alpha of 0.05 and power of  $0.8^{31}$ .





#### 6.2 Statistical Analysis:

The recorded simulation sessions will be reviewed by two separate pediatric emergency medicine and simulation experts who will evaluate the participants on the simulation global rating scale, a validated assessment tool for simulation. Inter-rater reliability will be calculated via Pearson correlation and ICC statistics, and the final reported value will be the mean of both reviewers.

The recorded sessions will also be reviewed to the time to metrics by two reviewers with a masked coinvestigator serving as the tie breaker in times of significant discordance. Time zero for the "time to" metrics will be when the facilitator finishes the scenario description.

The mean and 95% confidence interval of the metrics will be calculated for each group. Post randomization scores will be compared using a paired t-test, and with mixed effects linear models using pre-randomization score as a covariate. Time-to-event measures will be displayed with Kaplan Meier graphs and median time, and tested with the log-rank test, and secondarily using Cox proportional hazards models. Regression models may include adjustment for baseline variables imbalanced between arms or prognostic of outcome. Secondary Likert outcomes will be assessed with a proportional odds model. All results will be presented with appropriate 95% confidence intervals. Statistical analysis will be completed with statistician support using R statistical software.

#### **Protocol Deviations:**

All deviations will be reported to the REB in a timely manner.

#### 7 Data Handling and Record Keeping:

#### 7.1 Data Management Responsibilities:

The data will be stored on a secure redcap data-server. The server will be password protected and only the research team will have access to the data. Participant data will only be stored de-identified. The video recordings will be stored on an encrypted external hard drive kept in the PI's office locked office in a locked drawer. The original video data would be deleted from the simulation center.

#### 7.2 Record Retention

The data will be stored for 5 years after the publication of the study following which it will be destroyed. The data will be stored by BCCH.

#### 8 Budget & Finance:

Statistician and redcap access will be covered by the hospital/university due to being a fellow led project.

#### 9 Dissemination\Publication Plan:

Our knowledge translation plan includes manuscript publication in a peer-reviewed journal, and presentation at emergency medicine and/or pediatrics focused research conferences such as the PERC annual meeting.





#### 10 References:

- 1. Motola I, Devine LA, Chung HS, Sullivan JE, Issenberg SB. Simulation in healthcare education: A best evidence practical guide. AMEE Guide No. 82. *Medical Teacher*. 2013;35(10):e1511-e1530. doi:10.3109/0142159X.2013.818632
- 2. Kalnow A, Davis A, Hampton Z, Gable BD. In Situ Simulation to Promote Residents as Resuscitation Leaders. *Cureus*. 13(4):e14449. doi:10.7759/cureus.14449
- 3. Cook DA. If you teach them, they will learn: why medical education needs comparative effectiveness research. *Adv in Health Sci Educ*. 2012;17(3):305-310. doi:10.1007/s10459-012-9381-0
- 4. Johnston S, Coyer FM, Nash R. Kirkpatrick's Evaluation of Simulation and Debriefing in Health Care Education: A Systematic Review. *Journal of Nursing Education*. 2018;57(7):393-398. doi:10.3928/01484834-20180618-03
- 5. Zendejas B, Brydges R, Wang AT, Cook DA. Patient Outcomes in Simulation-Based Medical Education: A Systematic Review. *J Gen Intern Med.* 2013;28(8):1078-1089. doi:10.1007/s11606-012-2264-5
- 6. Okuda Y, Bryson EO, DeMaria Jr. S, et al. The Utility of Simulation in Medical Education: What Is the Evidence? *Mount Sinai Journal of Medicine*. 2009;76(4):330-343. doi:10.1002/msj.20127
- 7. Legoux C, Gerein R, Boutis K, Barrowman N, Plint A. Retention of Critical Procedural Skills After Simulation Training: A Systematic Review. *AEM Educ Train*. 2020;5(3):e10536. doi:10.1002/aet2.10536
- 8. Yang CW, Yen ZS, McGowan JE, et al. A systematic review of retention of adult advanced life support knowledge and skills in healthcare providers. *Resuscitation*. 2012;83(9):1055-1060. doi:10.1016/j.resuscitation.2012.02.027
- 9. Leigh G, Steuben F. Setting Learners up for Success: Presimulation and Prebriefing Strategies. *Teaching and Learning in Nursing*. 2018;13(3):185-189. doi:10.1016/j.teln.2018.03.004
- 10. Luctkar-Flude M, Tregunno D, Tyerman J, et al. Feasibility and Learning Outcomes Associated with Preparing Nursing Students for Simulation using Virtual Simulation Games. :1.
- 11. Drummond D, Delval P, Abdenouri S, et al. Serious game versus online course for pretraining medical students before a simulation-based mastery learning course on cardiopulmonary resuscitation: A randomised controlled study. *European Journal of Anaesthesiology* | *EJA*. 2017;34(12):836-844. doi:10.1097/EJA.0000000000000055
- 12. Bowyer MW, Hanson JL, Pimentel EA, et al. Teaching Breaking Bad News Using Mixed Reality Simulation. *Journal of Surgical Research*. 2010;159(1):462-467. doi:10.1016/j.jss.2009.04.032
- 13. Curtin LB, Finn LA, Czosnowski QA, Whitman CB, Cawley MJ. Computer-based Simulation Training to Improve Learning Outcomes in Mannequin-based Simulation Exercises. *AJPE*. 2011;75(6). doi:10.5688/ajpe756113





- 14. Franklin AE, Sideras S, Gubrud-Howe P, Lee CS. Comparison of Expert Modeling Versus Voice-Over PowerPoint Lecture and Presimulation Readings on Novice Nurses' Competence of Providing Care to Multiple Patients. *J Nurs Educ*. 2014;53(11):615-622. doi:10.3928/01484834-20141023-01
- 15. Mabry J, Lee E, Roberts T, Garrett R. Virtual Simulation to Increase Self-efficacy Through Deliberate Practice. *Nurse Educ*. 2020;45(4):202-205. doi:10.1097/NNE.0000000000000758
- 16. Moll-Khosrawi P, Zöllner C, Cencin N, Schulte-Uentrop L. Flipped learning enhances non-technical skill performance in simulation-based education: a randomised controlled trial. *BMC Medical Education*. 2021;21(1):353. doi:10.1186/s12909-021-02766-w
- 17. Tyerman J, Luctkar-Flude M, Graham L, Coffey S, Olsen-Lynch E. A Systematic Review of Health Care Presimulation Preparation and Briefing Effectiveness. *Clinical Simulation in Nursing*. 2019;27:12-25. doi:10.1016/j.ecns.2018.11.002
- 18. Tyerman J, Luctkar-Flude M, Graham L, Coffey S, Olsen-Lynch E. Pre-simulation preparation and briefing practices for healthcare professionals and students: a systematic review protocol. *JBI Database of Systematic Reviews and Implementation Reports*. 2016;14(8):80-89. doi:10.11124/JBISRIR-2016-003055
- 19. Birch L, Jones N, Doyle PM, et al. Obstetric skills drills: Evaluation of teaching methods. *Nurse Education Today*. 2007;27(8):915-922. doi:10.1016/j.nedt.2007.01.006
- 20. Zheng Z, Liao J, Zeng L, et al. High-Fidelity Patient Simulation Incorporated Into a Flipped Classroom Improves Students' Long-Term Knowledge Retention of Acute Organophosphorus Pesticide Poisoning. *Simulation in Healthcare*. 2022;17(1):e68. doi:10.1097/SIH.000000000000566
- 21. Blanie A, Shoaleh C, Marquion F, Benhamou D. Comparison of multimodal active learning and single-modality procedural simulation for central venous catheter insertion for incoming residents in anesthesiology: a prospective and randomized study. *BMC Medical Education*. 2022;22(1):357. doi:10.1186/s12909-022-03437-0
- 22. Stefaniak JE, Turkelson CL. Does the Sequence of Instruction Matter During Simulation? *Simulation in Healthcare: The Journal of the Society for Simulation in Healthcare*. 2014;9(1):15-20. doi:10.1097/SIH.0b013e3182a8336f
- 23. Zendejas B, Cook DA, Farley DR. Teaching First or Teaching Last: Does the Timing Matter in Simulation-Based Surgical Scenarios? *Journal of Surgical Education*. 2010;67(6):432-438. doi:10.1016/j.jsurg.2010.05.001
- 24. Thampi S, Lee CCM, Agrawal RV, et al. Ideal Sequence of Didactic Lectures and Simulation in Teaching Transesophageal Echocardiography Among Anesthesiologists. *Journal of Cardiothoracic and Vascular Anesthesia*. 2020;34(5):1244-1249. doi:10.1053/j.jvca.2019.12.011
- 25. Chua W, Burns R, Stone K, Reid J. Pediatric Emergency Medicine Simulation Curriculum: Hyponatremic Seizures. *MedEdPORTAL*. 12:10498. doi:10.15766/mep 2374-8265.10498





- 26. Friedman S, Tozzi M, Shakhin V, et al. Simulation of Seizures for the Pediatrics Resident. *MedEdPORTAL*. 10:9880. doi:10.15766/mep\_2374-8265.9880
- 27. Reid J, Stone K. Pediatric Emergency Medicine Simulation Curriculum: Seizure Scenario. *MedEdPORTAL*. 14:9794. doi:10.15766/mep 2374-8265.9794
- 28. Muir K, Buttle S, Shah M, trekk, EIIC. TREKK Pediatric Status Epilepticus Algorithm. Published online April 2022. Accessed September 30, 2022. https://trekk.ca/system/assets/assets/attachments/577/original/2022-05-02\_EIIC-Trekk Status Epilepticus Algorithm Final Version.pdf?1652215972
- 29. McKenzie KC, Hahn CD, Friedman JN, Canadian Paediatric Society Acute Care Committee. Emergency management of the paediatric patient with convulsive status epilepticus | Canadian Paediatric Society. CPS.ca. Published February 1, 2021. Accessed September 30, 2022. https://cps.ca/en/documents//position//emergency-management-of-the-paediatric-patient-with-convulsive-status-epilepticus/
- 30. Gaínza-Lein M, Sánchez Fernández I, Jackson M, et al. Association of Time to Treatment With Short-term Outcomes for Pediatric Patients With Refractory Convulsive Status Epilepticus. *JAMA Neurology*. 2018;75(4):410-418. doi:10.1001/jamaneurol.2017.4382
- 31. Kane S. Sample Size Calculator. ClinCalc.com. Published July 24, 2019. Accessed October 17, 2022. https://clincalc.com/stats/samplesize.aspx





## **Appendix A: Demographics:**

Please enter your age:

What is your experience with medical simulation?

a) No experience b) 1-5 simulation experiences c) 5-10 simulation experiences d) >10 simulation experiences

Before entering medicine please check any roles that apply?

- Background in ED Nursing
- Background as a paramedic or first responder?

#### **Confidence Quiz:**

Please rate your anxiety in the simulation experience from 1 to 5? 1 - Extremely anxious 5 - Not anxious at all

1 Extremely unknows 3 1vot unknows at an

Please rate your confidence in managing pediatric seizures in the future?

1 – Not confident at all, 5 – extremely confident

Please rate your satisfaction with the educational experience (Simulation + Debrief + Lecture)?

 $1-extremely\ dissatisfied\ ,\ 5\ extremely\ satisfied$ 





#### Appendix B



#### Case Presentation

You are working in the ED and a 4 year old girl is brought in who has been having generalized tonic-clonic movements and head deviation for the past 10 minutes.

- What is the diagnosis?
- What might be the underlying cause?
- How do you stabilize this patient?
- What's the best way to stop this seizure?
- Are there any tests or investigations you need to think about?

#### What is status Epilepticus?





# Differential for Seizures Important aspects to consider: • EMS handover • SAMPLE History: • Signs & Symptoms • Fever • head injuries • Allergies • Medications • Taking • Medication at home • Past Medical History • Last meal • Events leading up to presentation











#### Stabilization

#### Initial Management

- Initiate ABCs, cardiorespiratory and BP monitoring

  0, 10-15 L/min via non-rebreather mask
  Prioritize giving the first dose of benzodiazepine as early as possible, followed by checking blood glucose
  Monitor for respiratory depression, hypotension, arrhythmias
  Give acetaminophen 15 mg/kg/dose [MAX 650 mg] PR if febrile

- Consider other investigations:
  Electrolytes, blood gas, calcium, CBC, serum glucose
  Other: anticonvulsant drug levels, LFTs, blood & urine culture

#### Primary Survey - A - Airway





#### Primary Survey - B - Breathing



#### Primary Survey - C - Circulation





#### Primary Survey - D - Disability







#### Primary Survey - E - Exposure



#### Estimating your patients weight





#### First line Treatment































#### Raised ICP/Trauma/Stroke

Necessary Investigations:
Non-Contrast CT Scan

- Band-Aids:
  Head of bed elevation
  Sedation
  Hypertonic saline
  Mannitol
  Hyperventilation

- Managing secondary brain injury:
  Normothermia
  Normotension
  Normoglycemia





#### Infection

- Febrile Seiture:

  Between 6 months and 6 year with a temp >38.0C

  Absence of CNS infection/inflammation and no acute systemic abnormalities

  Seizures typically 5-10 mins with shorter post-ictal period of 5-10 mins.

- Febrile Status Epilepticus Consider Meningitis/Encephalitis Blood Culture Urine Culture Consider LP/CSF if stable

Start antibiotics as soon as possible





#### Disposition

- Discharging:

  Ensure neurology follow up

  Outpatient EEG

  +/- Outpatient MRI

Brief Febrile Seizure - No further investigations needed

# Admission Investigations: Neurology Consult MRI Brain Lumbar Puncture EEG Metabolic Workup



#### Resources









#### References

- (2021) Twitter. Metrolina Trauma Advisory Committee, 30 August. Available at: https://twitter.com/metrolinatrauma/status/1432353465758531588 (Accessed: January 12, 2023).
- Gary Heiting, O.D. (2019) Dilated pupils: Causes and concerns, All About Vision. All About Vision. Available at: https://www.allaboutvision.com/conditions/dilated-pupils.htm (Accessed: January 12, 2023).
- Libod, G. (2021) sist rinnyy mang-aneticky, ECML enter Rys, Analble et Intra/Jowaccement/#15x819573195 (ed. 1874). Analble et Intra/Jowaccement/#15x81957319519-ffel8f4-1a10 (Accessed: January 11, 2023). Areabon shylinic arm (no date) Steparior. Analble et Intra/Jowaccement/#15x81957319519-ffel8f4-1a10 (Accessed: January 12, 2023). A Feebron shylinic arm (no date) Steparior. Analble et Intra/Jowaccement/#15x919-ffel8f4-1a10 (Accessed: January 12, 2023). Strider: Lang Sounds: MEDICADO (10218) YouTube. VouTube. Available at: https://www.youtube.com/watch?v=5dE(79146w/kccessed: January 11, 2023).
- (Accessed: January 11, 2023).

  Chua W, Burra R, Stone K, Red J. Pediatric Emergency Medicine Simulation Curriculum: Hyponatremic Seitures. MedIdPORTAL. 1210486. doi:10.1756/jmlep\_1274-8265.10488

  Friedmans, Tozzi M, Dabahn V, et al. Simulation of Seitures for the Pediatrics Resident. MedIdPORTAL. 103880. doi:10.1046/jmlep\_1274-8265.5048
- Reid J, Stone K, Pediatric Emergency Medicine Simulation Curriculum: Seizure Scenario. MedEdPORTAL. 14:9794.
  doi:10.15766/mep. 2374-8265-39794 GOI: JLI-J7-00/Imp\_\_z3/4-20-3/394
  Mulir K, Buttle S, Shah M, Yrekk EllC TREKK Pediatric Status Epilepticus Algorithm. Published online April 2022. Acc
  30, 2022. https://trekk.ca/system/assets/assets/attachments/S77/original/2022-05-02\_EllCTrekk Status\_Epilepticus\_Algorithm=final\_Version\_orpf?165221236.
- McKenzie KC, Hahn CD, Friedman JN, Canadian Paediatric Society Acute Care Committee. Emergency management of the paediatric patient with convulsive status epilepticus | Canadian Paediatric Society. CPS.ca. Published February 1, 2021. Accessed September 30, 2022. https://cps.ca/en/documents//position//emergency-management-of-the-paediatric-patient-with-convulsive-status-epilepticus/





The quiz answers will be available at the end of the study should you be interested





Guidelines: ⊠ Appendix B

Flowsheets:

Appendix C Scenario 1 Case Title: Status epilepticus in an 8-year-old child **Author:** John Ramsay

Date Last Updated: 2022-11-30 Reason for Development: Simulation research scenario **Target Population:** 2<sup>nd</sup> year medical students Target Duration: 10 minute simulation **Learning Objectives:** 1. ABC approach in a sick child 2. Initiation of seizure management and review of Trekk Algorithm 3. Initiation of basic seizure investigations **Core Competencies Checklist:** Medical Expert: ⊠ Professional: ⊠ Communicator: ⊠ Collaborator: □ Leader: ⊠ Health Advocate: □ Scholar: □ **Crisis Resource Management Skills:** Know Environment: ⊠ Anticipate & Plan: ⊠ Call for help early: ⊠ Distribute workload: □ Exercise leadership & Followership: □ Mobilize all available resources: ☐ Use all information: ⊠ Re-evaluate case: ⊠ Prevent & Manage Fixation errors: □ Use good teamwork: ⊠ Communicate effectively:  $\boxtimes$  Allocate attention:  $\boxtimes$  Set priorities dynamically  $\boxtimes$ **Scenario Setup: Clinical Setting:** ED Resus Room: Sim Lab: ⊠ Other: \( \sum \) Ward Low fi infant: □ Low-fi Child: ⊠ High-Fi Infant: □ High-fi Child: ⊠ System: **Equipment Needs:** ☐ Airway cart (Laryngoscope, ETT, etc) ☐ Chest tube set up  $\bowtie$  Bed ☐ Three-way stopcock ⊠Medication Cart ☐ Foley Catheter  $\square$  IV Pump + Pole ⊠ Vitals: chest leads, pulse ox, Bp cuff ☐ Defibrillator/Pacer/ECG Leads  $\square$  PPE ⊠ O<sub>2</sub> delivery (NP, NRB mask, BVM) ☐ IO Setup **Adjuncts Needed:** 

Bloodwork: ⊠ Appendix A

Videos/Photos: □

Protocol number: 1 Version date: 16-Aug-23

ECG: □

Imaging: □

Page 18 of 27





Age: 8 yrs Sex: Male Wt: 30kg

#### **Case Summary (For Facilitator):**

8-year-old male presenting to the ED who has been having seizure for the past 10 minutes. His seizures will resolve following the administration of a second line anti-epileptic. The scenario is complicated by inability to obtain IV access for the first dose and worsening airway protection and desaturation as the case progresses. IV access can be obtained after an initial intranasal dose of midazolam is given.

#### Case Intro/Clinical Vignette (Read out loud to participants):

The paramedics are about to arrive with Rahul an 8-year-old male who is unresponsive and has been having tonic-clonic movements of his limbs for the past 10 minutes.

#### **Additional Hx** (if asked):

HPI: previous well

PMH: Nil Meds: Nil Algs: Nil





Stage 1:

| Patient Condition | Simulator<br>Parameters | Effective Management | Consequences of ineffective management | Notes: |
|---|---|---|---|---|
| General: Unresponsive, no work of breathing, normal colour Airway: No stridor, neck flexed, Breathing: No WOB, normal chest rise Circulation: Normal pulses, cap refill <3, warm extremities | HR: 122<br>RR: 10<br>SaO <sub>2</sub> : 90%<br>BP: 110/75<br>Temp: 37.7C | A: • Attempt better positioning • Jaw thrust • Suction • Oral Airway | | IV access is<br>unsuccessful |
| <b>Disability:</b> Unresponsive, Pupils dilated, reactive | | B: O <sub>2</sub> by non-rebreather or | | |
| P/E: Cardio: Unremarkable Resp: Unremarkable Abdo: unremarkable | | facemask C: • Attempt IV access | | |
| Neuro: Pupils dilated, no reflexes,<br>stiff tone, repeated flexion of arms,<br>head deviation to one side | | • Cycle BP's Monitors: | | |
| | | Chest leads, sat monitor, BP Cuff | | |
| | | Investigations: • POC Glucose (4.0) • Blood work | | |





| Medications: |
|---------------------------------------------------------|
| <ul> <li>Intranasal Midaz<br/>or Diazepam PR</li> </ul> |
| or biazepain PK |

Stage 2:

| Patient Condition | Simulator Parameters | Effective Management | Consequences of ineffective management | Notes: |
|---|---|---|---|---|
| General: 5 minutes have passed, and patient is continuing to seize Airway: No intervention: Mild stridor, poor position Intervention: supported effectively Breathing: If no jaw thrust mild work of breathing, otherwise unremarkable Circulation: Normal pulses, normal cap refill Disability: Unresponsive | HR: 126 RR: 12 SaO <sub>2</sub> : 84% if no intervention 95 if O <sub>2</sub> and airway management BP: 112/80 Temp: 37.8 | A: | Need to get to second line agent to abort seizure | |
| P/E: Unchanged | | | | |

| Expected / Critical Actions | Unacceptable Actions: |
|---|---|
| Attempted IV access and repeat attempt later | No airway management when patient is stridulous |





- Transition to Non-IV medication when access unavailable
- Call for support (Neuro) if seizure continues

#### **Medical Expert Points to bring up for discussion:**

- Intranasal midazolam vs IV Lorazepam and effectiveness
- Importance of airway management
- Work-up for unknown seizure (Glucose, lytes)

| Lab | Result | Normal Range |
|---|---|---|
| CBC | | |
| WBC | 7 x 10 <sup>9</sup> | 4-12x10 <sup>9</sup> |
| Hgb | 130 | 130 – 160 |
| Plt | 320 | 150 – 450 |
| Glucose | 5.7 | |
| Electrolytes & Extended electrolytes: | | |
| Sodium (Na <sup>+</sup> ) | 140 | 135 – 145 |
| Potassium (K <sup>+</sup> ) | 4.2 | 3.5 – 5.5 |
| Chloride (Cl <sup>-</sup> ) | 103 | 102 – 112 |
| Ionized Calcium (iCa) | 1.18 | 1.15 – 1.3 |
| Phosphate (PO4 <sup>-2</sup> ) | 1.5 | 1.16 – 1.81 |
| Magnesium (Mg <sup>2+</sup> ) | 0.8 | 0.66 – 0.91 |





| Scenario 2 | | | | |
|---|---|---|---|---|
| Case Title: Status e | pilepticus in a 1-year-old child | | Author: John Ramsay | Date Last Updated: 2022-11-30 |
| | pment: Simulation research scenar | io | | |
| | 2 <sup>nd</sup> year medical students | | | |
| | 0 minute simulation | | | |
| Learning Objective | | | | |
| 1. ABC approach ir | n a sick child | | | |
| 2. Initiation of seiz | ure management and review of Tre | ekk Algorithm | | |
| 3. Initiation of bas | ic seizure investigations | | | |
| Cana Cammatamaia | s Charliste | | | |
| Core Competencie | | ✓ Callahamatam ☐ I a | adam M. Haalth Advanata. | Scholar: □ |
| Crisis Resource M | Professional: Communicator: | △ Conaborator: ☐ Lea | ader: 🖂 Health Advocate: 🗆 | Scholar: |
| | anagement Skins:<br>: ⊠ Anticipate & Plan: ⊠ Call f | or halm apply: \(\sime\) Distribu | ta wanklaadi 🗆 Evaraisa laa | darshin & Fallayyarshin, |
| | le resources: Use all information | - · | | - |
| | | | _ | e Fixation errors: $\square$ Use good teamwork: $\boxtimes$ |
| | tively: Allocate attention: S | Set priorities dynamically | × | |
| Scenario Setup: | | C: I 1 🖂 | 0.1 | |
| Clinical Setting: | ED Resus Room: | Sim Lab: ⊠ | Other: Ward | TT 1 0 01 11 1 |
| System: | Low fi infant: $\square$ | Low-fi Child: □ | High-Fi Infant: 🗵 | High-fi Child: □ |
| <b>Equipment Needs:</b> | | | | |
| ⊠ Bed | | ☐ Airway cart (Laryng | goscope, ETT, etc) | ☐ Chest tube set up |
| ⊠Medication Cart | | | | ☐ Three-way stopcock |
| $\square$ IV Pump + Pole | | | oulse ox, Bp cuff | ☐ Foley Catheter |
| ☐ Defibrillator/Pac | er/ECG Leads | $\square$ PPE | | |
| $\boxtimes$ O <sub>2</sub> delivery (NP, | NRB mask, BVM) | ☐ IO Setup | | |
| <b>Adjuncts Needed:</b> | • | - | | |
| ECG: □ | | Bloodwork: Apper | ndix A | Guidelines: Appendix B |
| Imaging: □ | | Videos/Photos: □ | | Flowsheets: |

Protocol number: 1 Version date: 16-Aug-23 Page 23 of 27





Age: 1 yr Sex: Female Wt: 10kg

#### **Case Summary (For Facilitator):**

1-year-old girl presenting on the ward who has been having seizure for the past 5 minutes. Her seizures will resolve following the administration of a second line anti-epileptic. The scenario is complicated by inability to obtain IV access for the first dose and worsening airway protection and desaturation as the case progresses. IV access can be obtained after an initial intranasal dose of midazolam is given.

#### **Case Intro/Clinical Vignette (Read out loud to participants):**

The nurse calls you about with Zoe a 1-year-old girl who is unresponsive and has been having tonic-clonic movements of her limbs for the past 5 minutes. She was admitted for gastroenteritis and pulled her IV out earlier today.

#### **Additional Hx** (if asked):

HPI: previous well

PMH: Nil Meds: Nil Algs: Nil





## Stage 1:

| Patient Condition | Simulator<br>Parameters | Effective Management | Consequences of ineffective management | Notes: |
|---|---|---|---|---|
| General: Unresponsive, no work of breathing, normal colour Airway: No stridor, neck flexed, Breathing: No WOB, normal chest rise Circulation: Normal pulses, cap refill <3, warm extremities Disability: Unresponsive, Pupils dilated, reactive P/E: Cardio: Unremarkable Resp: Unremarkable Abdo: unremarkable Neuro: Pupils dilated but reactive,, no reflexes, stiff tone, repeated flexion of arms, head deviation to one side | HR: 170<br>RR: 14<br>SaO₂: 90%<br>BP: 95/55<br>Temp: 37.6C | A: Attempt better positioning Jaw thrust Suction Oral Airway B: O <sub>2</sub> by non-rebreather or facemask C: Attempt IV access Cycle BP's Monitors: Chest leads, sat monitor, BP Cuff Investigations: POC Glucose (2.0) Blood work Medications: Intranasal Midaz or Diazepam PR Call for help | | IV access is<br>unsuccessful |





Stage 2:

| Patient Condition | Simulator Parameters | Effective Management | Consequences of ineffective management | Notes: |
|---|---|---|---|---|
| General: 5 minutes have passed, and patient is continuing to seize Airway: No intervention: Mild stridor, poor position Intervention: supported effectively Breathing: If no jaw thrust mild work of breathing, otherwise unremarkable Circulation: Normal pulses, normal cap refill Disability: Unresponsive P/E: Unchanged | HR: 126 RR: 12 SaO <sub>2</sub> : 84% if no intervention 95 if O <sub>2</sub> and airway management BP: 112/80 Temp: 37.8 | A: | <ul> <li>Need to get to second line agent to abort seizure</li> <li>Should correct glucose to stop seizure.</li> </ul> | |

| Expected / Critical Actions | Unacceptable Actions: |
|---|---|
| Attempted IV access and repeat attempt later | <ul> <li>No airway management when patient is stridulous</li> </ul> |
| <ul> <li>Transition to Non-IV medication when access</li> </ul> | |
| unavailable | |
| Call for support (Neuro/Staff) if seizure continues | |

#### **Medical Expert Points to bring up for discussion:**

- Intranasal midazolam vs IV Lorazepam and effectiveness
- Importance of airway management
- Work-up for unknown seizure (Glucose, lytes)





| Lab | Result | Normal Range |
|--------------------------------|---------------------|----------------------|
| СВС | | |
| WBC | 8 x 10 <sup>9</sup> | 4-12x10 <sup>9</sup> |
| Hgb | 145 | 130 – 160 |
| Plt | 270 | 150 – 450 |
| Glucose | 4.2 | |
| Electrolytes & Extended | | |
| electrolytes: | | |
| Sodium (Na <sup>+</sup> ) | 144 | 135 – 145 |
| Potassium (K <sup>+</sup> ) | 4.5 | 3.5 – 5.5 |
| Chloride (Cl <sup>-</sup> ) | 103 | 102 – 112 |
| Ionized Calcium (iCa) | 1.2 | 1.15 – 1.3 |
| Phosphate (PO4 <sup>-2</sup> ) | 1.4 | 1.16 - 1.81 |
| Magnesium (Mg <sup>2+</sup> ) | 0.8 | 0.66 - 0.91 |